CLINICAL TRIAL: NCT05644366
Title: Proprioception and Vestibular Alterations Affect Postural Control in Children With Mild Autism: A Pilot Study
Brief Title: Postural Control Instability in Children With Mild Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: A2540214
Record Dates: First submitted 2018-02-28; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The balance assessment procedure included the following; each subject was instructed to stand on both feet for 15 seconds on the pressure MatScan under eight different conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Balance Assessment Children with Autism (Experimental): Postural Stability Testing Each subject was instructed to stand in a static bipedal posture on the MatScan® pressure mat and performed 8 balance tasks.
  Interventions: Other: Postural Control Balance Assessment

INTERVENTIONS:
Other: Postural Control Balance Assessment — Postural Stability Testing Each subject was instructed to stand in a static bipedal posture on the MatScan® pressure mat and performed 8 balance tasks.

SUMMARY:
Objective: Individuals diagnosed with Autism Spectrum Disorder (ASD) exhibit some type of motor control impairment, for instance, motor apraxia and history of gross motor delay that could lead to increased risk of fall. This pilot research was designed to assess and characterize static postural stability and create a starting point to better understand and describe postural control in children with mild autism. Method: We measured static postural control with center of pressure (COP) displacement in 10 children with mild autism during eight sensory conditions that challenge and cancel the visual, proprioceptive and vestibular systems.

DETAILED DESCRIPTION:
Materials and methods Institutional Review Board (IRB) approval at the University of Puerto Rico, Medical Science Campus has obtained prior the recruitment of the participants. Parents of children diagnosed with mild ASD who were interested in the study called the number on the recruitment flyer. The PI spoke with the parent to assess whether their child qualified for the study based on the following inclusion and exclusion criteria.

Balance Assessment Protocol

The balance assessment procedure included the following; each subject was instructed to stand on both feet for 15 seconds on the pressure MatScan under eight different conditions. The first four conditions were executed over a stable surface and consisted of the following: (1) eyes open (EO) -evaluates visual, vestibular and proprioceptive systems, (2) eyes closed (EC) -eliminates visual input, evaluates vestibular and proprioceptive system, (3) eyes open while moving head up and down (at 60 beats per minute) (EO HUD) -evaluates visual and proprioceptive system and alters vestibular input, (4) eyes closed while moving the head up and down (EC HUD) -evaluates the effect of removing visual information, and the vestibular input being altered. The subjects then performed the same four tasks, this time standing on an unstable platform (high quality closed cell foam 19 inches long x 15 inches width x 2.25 inches)with the purpose of altering the proprioceptive input and increasing dependence on the visual and vestibular systems.

ELIGIBILITY:
Inclusion Criteria:

* children from 7-12 years of age, male or female
* mild ASD diagnosis (as determined by a medical doctor)
* capable of ambulating independently.

Exclusion Criteria:

* children with additional neurological problems
* children with visual problems
* children unable to tolerate walking or standing barefoot
* children who have fallen three or more times in the last three months
* children with vestibular problems.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2014-08-14 (Actual); Primary Completion 2015-08-14 (Actual); Study Completion 2015-09-14 (Actual)

PRIMARY OUTCOMES:
Postural Stability | Baseline
  Postural stability was operationally defined by the center of pressure displacement measured by the MatScan® pressure mat. These sensors detect the displacement as the body sways anterior, posterior or laterally (right or left).

CONTACTS AND LOCATIONS:
Overall Officials: Martin G. Rosario, PT, PhD, Principal Investigator — Texas Woman's University

REFERENCES:
- [Background] Ming X, Brimacombe M, Wagner GC. Prevalence of motor impairment in autism spectrum disorders. Brain Dev. 2007 Oct;29(9):565-70. doi: 10.1016/j.braindev.2007.03.002. Epub 2007 Apr 30. PMID 17467940
- [Background] Teitelbaum P, Teitelbaum O, Nye J, Fryman J, Maurer RG. Movement analysis in infancy may be useful for early diagnosis of autism. Proc Natl Acad Sci U S A. 1998 Nov 10;95(23):13982-7. doi: 10.1073/pnas.95.23.13982. PMID 9811912
- [Background] Fournier KA, Kimberg CI, Radonovich KJ, Tillman MD, Chow JW, Lewis MH, Bodfish JW, Hass CJ. Decreased static and dynamic postural control in children with autism spectrum disorders. Gait Posture. 2010 May;32(1):6-9. doi: 10.1016/j.gaitpost.2010.02.007. Epub 2010 Apr 18. PMID 20400311
- [Background] Mari M, Castiello U, Marks D, Marraffa C, Prior M. The reach-to-grasp movement in children with autism spectrum disorder. Philos Trans R Soc Lond B Biol Sci. 2003 Feb 28;358(1430):393-403. doi: 10.1098/rstb.2002.1205. PMID 12639336
- [Background] Kohen-Raz R, Volkmar FR, Cohen DJ. Postural control in children with autism. J Autism Dev Disord. 1992 Sep;22(3):419-32. doi: 10.1007/BF01048244. PMID 1383190
- [Background] Fournier KA, Hass CJ, Naik SK, Lodha N, Cauraugh JH. Motor coordination in autism spectrum disorders: a synthesis and meta-analysis. J Autism Dev Disord. 2010 Oct;40(10):1227-40. doi: 10.1007/s10803-010-0981-3. PMID 20195737
- [Background] Blanche EI, Reinoso G, Chang MC, Bodison S. Proprioceptive processing difficulties among children with autism spectrum disorders and developmental disabilities. Am J Occup Ther. 2012 Sep-Oct;66(5):621-4. doi: 10.5014/ajot.2012.004234. PMID 22917129
- [Background] Shumway-Cook, A., & Woollacott, M. H. (2001a). Constraints of motor control. Motor control: Theory and practical applications (2nd ed., pp. 127-161). Philadelphia, Pa. ; London: Lippincott Williams & Wilkins.
- [Background] Kern, J. K., Garver, C. R., Grannemann, B. D., Trivedi, M. H., Carmody, T., Andrews, A. A., & Mehta, J. A. (2007). Response to vestibular sensory events in autism. Research in Autism Spectrum Disorders, 1(1), 67-74. doi:10.1016/j.rasd.2006.07.006
- [Background] Molloy CA, Dietrich KN, Bhattacharya A. Postural stability in children with autism spectrum disorder. J Autism Dev Disord. 2003 Dec;33(6):643-52. doi: 10.1023/b:jadd.0000006001.00667.4c. PMID 14714933
- [Background] Shumway-Cook, A., & Woollacott, M. H. (2001b). Development of postural control. Motor control: Theory and practical applications (2nd ed., pp. 192-221). Philadelphia, Pa. ; London: Lippincott Williams & Wilkins.
- [Background] FUKUDA T. The stepping test: two phases of the labyrinthine reflex. Acta Otolaryngol. 1959 Mar-Apr;50(2):95-108. doi: 10.3109/00016485909129172. No abstract available. PMID 13636842
- [Background] Zammit GV, Menz HB, Munteanu SE. Reliability of the TekScan MatScan(R) system for the measurement of plantar forces and pressures during barefoot level walking in healthy adults. J Foot Ankle Res. 2010 Jun 18;3:11. doi: 10.1186/1757-1146-3-11. PMID 20565812
- [Background] Hansson EE, Beckman A, Hakansson A. Effect of vision, proprioception, and the position of the vestibular organ on postural sway. Acta Otolaryngol. 2010 Dec;130(12):1358-63. doi: 10.3109/00016489.2010.498024. Epub 2010 Jul 16. PMID 20632903
- [Background] O'sullivan, S. B. (2007). Examination of motor function: Motor control and motor learning. Physical rehabilitation (pp. 233-234) FA Davis Company Philadelphia.